CLINICAL TRIAL: NCT03400670
Title: Comparison of Two Different NCPAP Methods in Preterm Infants With Respiratory Distress Syndrome With Gestational Age of 26-30 Weeks
Brief Title: Comparison of Two Different NCPAP Methods in Preterm Infants With Respiratory Distress Syndrome
Acronym: (NCPAP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02082019
Record Dates: First submitted 2017-12-11; First posted 2018-01-17 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2017-01

CONDITIONS: Ventilatory Failure
Keywords: NCPAP; Respiratory Distress Syndrome
MeSH Terms: conditions — Hypoventilation; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilator NCPAP (Active Comparator): neonatal ventilator (SLE; Specialised Laboratory Equipment, UK) PEEP: 5 cmH2O
  Interventions: Device: ventilator NCPAP
- Infant Flow-driver NCPAP (Active Comparator): infant flow-driver device (Infant Flow System, Viasys Corp., USA) PEEP:5-8 cmH2O, This group receive variable flow
  Interventions: Device: ventilator NCPAP

INTERVENTIONS:
Device: ventilator NCPAP — infants will be randomized into two different NCPAP groups
  Other Names: infant flow driver NCPAP

SUMMARY:
is to compare introduction of two different NCPAP methods in terms of mechanical ventilation (MV) need (non-invasive respiratory support failure) and surfactant need within the first 72 hours of life in preterm infants with Respiratory Distress Syndrome (RDS) at 26-30 weeks of gestation.

DETAILED DESCRIPTION:
Study Design NCPAP support was provided with continuous positive airway pressure, which was generated by a neonatal ventilator (SLE; Infant Flow System, Viasys Corp., USA) and infant flow-driver device (SLE; The respiratory parameter settings were a PEEP of 5-8 cmH2O. CPAP was stopped when PEEP 5 cmH2O and infants showed no signs of RDS with FiO2 <0.30.

Under non-invasive respiratory support, in case of FiO2 is ≥ 0.40, surfactant will be given as early rescue therapy by means of non-invasive method (by using a thin catheter - take care method- while spontaneous breathing continues) in order to keep target oxygen saturation between 90-95 %. The second dose of surfactant will be given 6 hours after the first dose by means on non-invasive method in order to keep target oxygen saturation between 90-95 % in case of FiO2 need is ≥ 0.30.

Non-invasive respiratory support failure is set as follows:

* FiO2 of ≥ 0.50 in order to keep oxygen saturation measured by pulse oximetry above 90 % and higher,
* Apnea requiring more than 6 alerts in a 24 -hour period in 6 consecutive hours or more than 1 apnea requiring positive pressure ventilation,
* Persistent acidosis; presence of pH < 7.20 and PCO2 > 65 mmHg in two different blood gases drawn with an interval of at least 30 minutes or treatment-resistant metabolic acidosis,
* Severe respiratory distress,
* Pulmonary haemorrhage and cardiopulmonary arrest.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant with gestational age of 26 weeks 0 days and 29 weeks 6 days with RDS signs will be included

Exclusion Criteria:

* Major congenital anomalies
* Presence of cardiovascular instability
* Intubation at admission to the NICU
* Consent not provided or refused

Ages: 1 Hour to 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2017-01-05 (Actual); Primary Completion 2020-01-05 (Estimated); Study Completion 2020-02-05 (Estimated)

PRIMARY OUTCOMES:
noninvasive ventilation failure | 72 hours
  need for mechanical ventilation in the first 72 hours of life

CONTACTS AND LOCATIONS:
Overall Officials: Suna Oğuz, Study Director — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Maternity Teaching, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No